CLINICAL TRIAL: NCT01903551
Title: Phase 3 Study of Post-operative Pain Management With Loco-regional Analgesia in Minithoracotomy for Cardiac Surgery. A Randomized Controlled Trial
Brief Title: Loco-regional Analgesia for Post-operative Pain Management in Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Daniela Pasero, Medical Doctor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTurin
Record Dates: First submitted 2013-07-13; First posted 2013-07-19 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Pain, Postoperative
Keywords: post-operative pain; loco-regional analgesia; minimally invasive surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loco-regional catheter (Experimental): A suprafascial catheter will be positioned at the end of cardiac intervention during the thoracotomy closure. The catheter will be connected to a elastomeric pump, which delivers the analgesic drug (ropivacaine).
  Interventions: Device: Loco-regional catheter
- Intravenous analgesia (No Intervention): At the end of the cardiac intervention each patient will receive intravenous analgesia with morphine at 0.8 mg/h.

INTERVENTIONS:
Device: Loco-regional catheter — it is an intra-fascial catheter for realing of the drug locally
  Arms: Loco-regional catheter

SUMMARY:
The aim of the study is to evaluate whether loco-regional analgesia reduces post operative pain compared to intravenous analgesia, in patients undergoing cardiac surgery in minithoracotomy. All patients will be randomized to receive locoregional analgesia (treatment group) or intravenous analgesia (control group), at the end of the cardiac intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing minithoracotomy for cardiac surgery, > 18 years old

Exclusion Criteria:

* psychiatric diseases, which might limit pain evaluation; urgent surgery; patients on ECMO; lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
ICU lenght of stay and hospital stay | 28 days

SECONDARY OUTCOMES:
Mechanical ventilation in the post-operative period | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiac Intensive Care Unit, Turin, Italy, Italy